CLINICAL TRIAL: NCT06486480
Title: Effect of Minimally Invasive Surgical Assisted by Robots on Intraventricular Hemorrhage
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jin Hu (Other)
Responsible Party: Sponsor-Investigator, Jin Hu, Huashan Hospital, Fudan University, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSSJWK202406
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Clarify the Therapeutic Differences Between Robot Assisted Endoscopic Clearance and Traditional Puncture and External Drainag

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted endoscopy group (Experimental): Using robot assisted endoscopy to clear intraventricular hemorrhage
  Interventions: Procedure: Using robot assisted endoscopy to clear intraventricular hemorrhage
- External ventricular drainage group (Active Comparator): Using External ventricular drainage to clear intraventricular hemorrhage
  Interventions: Procedure: Using robot assisted endoscopy to clear intraventricular hemorrhage

INTERVENTIONS:
Procedure: Using robot assisted endoscopy to clear intraventricular hemorrhage — More advanced surgical auxiliary instruments are used to improve surgical accuracy
  Other Names: External ventricular drainage

SUMMARY:
Clarify the therapeutic differences between robot assisted endoscopic clearance and traditional puncture and external drainage, and establish a new minimally invasive surgical diagnosis and treatment strategy for intraventricular hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 80 years old;

  * The time from onset to first CT confirmation of intraventricular hemorrhage is less than 24 hours;

    * Before enrollment, CT confirmed that the intraventricular hemorrhage score (modified Graeb score) was ≥ 8 points, and the total score of bilateral lateral ventricles was ≥ 5 points;

      * If there is concurrent cerebral hemorrhage but the hematoma volume is less than 30ml;

        ⑤ First CT to surgery time<72 hours;

        ⑥ GCS ≤ 14.

Exclusion Criteria:

* ① Suspected (unless excluded by angiography or CTA/MRA/MRI) or untreated rupture of cerebral aneurysm, Moyamoya disease, intracranial AVM rupture, or tumor;

  * Patients with a GCS score of 3 and/or fixed dilated pupils and/or no spontaneous breathing;

    * Patients with pre-existing neurological disorders that affect neurological function assessment prior to onset;

      * Coagulation dysfunction;

        * Patients who require long-term anticoagulant treatment;

          ⑥ Use dabigatran, apixaban, and/or rivaroxaban (or drugs of the same class) before symptoms appear; ⑦ Platelet count<100 × 109/L, INR>1.4;

          ⑧ Pregnancy (positive serum or urine pregnancy test);

          ⑨ Subtentorial hemorrhage or brainstem hemorrhage;

          ⑩ Patients who have previously participated in other interventional clinical studies and participated in observational, natural history, and/or epidemiological studies that do not involve intervention are eligible;

          ⑪ Subjects who are expected to not survive until the 180th day of visit; No written informed consent was given by the subjects or legal representatives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month mRS score | 180 days
  MRS Scores 6 months after onset

SECONDARY OUTCOMES:
30 day mortality rate | 0-30 days
  Mortality at 30 days after onset